CLINICAL TRIAL: NCT03504423
Title: A Phase III Multicenter Open-label Randomized Trial to Evaluate Efficacy and Safety of Folfirinox (FFX) Versus Combination of CPI-613 With Modified Folfirinox (mFFX) in Patients With Metastatic Adenocarcinoma of the Pancreas
Brief Title: Study Evaluating Efficacy and Safety of FFX Versus Combination of CPI-613 With mFFX in Patients With Metastatic Adenocarcinoma of the Pancreas
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cornerstone Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PANC003
Record Dates: First submitted 2018-04-12; First posted 2018-04-20 (Actual); Results first posted 2023-01-03 (Actual); Last update posted 2023-01-03 (Actual); Status verified 2021-09

CONDITIONS: Pancreatic Cancer Metastatic
MeSH Terms: interventions — devimistat; Leucovorin; Irinotecan; folfirinox; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CPI-613, mFolfirinox (Experimental): CPI-613, mFolfirinox
  CPI-613 at 500 mg/m2 IV infusion at a rate of 4mL/min via a central venous port on day 1 and 3 of a 14-day cycle.
  mFolfirinox (given immediately after CPI-613 administration): Oxaliplatin (Eloxatin) at 65 mg/m2 given as a 2 hr IV infusion, Folinic acid at 400 mg/m2 given as a 90 min (1.5hr) infusion immediately after Oxaliplatin, and concurrently with Irinotecan (irinotecan at 140mg/m2 given as a 90 min IV infusion) via a Y-connector, Flurouracil at 400 mg/m2 as bolus followed by a 46 hr infusion at 2400mg/m2 starting immediately after completion of folinic acid and Irinotecan.
  Interventions: Drug: CPI 613, mFolfirinox
- Folfirinox (Active Comparator): Folfirinox
  Folfirinox: Oxaliplatin (Eloxatin) at 85 mg/m2 given as a 2 hr IV infusion, Folinic acid at 400 mg/m2 given as a 90 min (1.5hr) infusion immediately after Oxaliplatin, and concurrently with Irinotecan (irinotecan at 180mg/m2 given as a 90 min IV infusion) via a Y-connector, Flurouracil at 400 mg/m2 as bolus followed by a 46 hr infusion at 2400mg/m2 starting immediately after completion of folinic acid and Irinotecan.
  Interventions: Drug: Folfirinox

INTERVENTIONS:
Drug: CPI 613, mFolfirinox — CPI-613: 500mg/m2, IV infusion at a rate of 4mL/min via a central venous port. mFolfirinox: given immediately after CPI-613 administration
  Other Names: CPI-613,Oxaliplatin, folinic acid, irinotecan, flurouracil
  Arms: CPI-613, mFolfirinox
Drug: Folfirinox — Folfirinox
  Other Names: Oxaliplatin, folinic acid, irinotecan, flurouracil
  Arms: Folfirinox

SUMMARY:
A prospective, multicenter, open label, randomized phase III study to evaluate efficacy and safety of FFX versus CPI-613 + mFFX in patients with metastatic adenocarcinoma of the pancreas with age range of 18 to 75 years

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed metastatic Stage IV adenocarcinoma of the pancreas
2. No prior treatments for stage IV pancreatic adenocarcinoma (prior adjuvant or neoadjuvant treatment is allowed provided completed > 6 months prior to disease recurrence)
3. Eastern Cooperative Oncology Group (ECOG) performance status 0 - 1
4. Male and female patients 18 - 75 years of age
5. Measurable disease determined using guidelines of Response Evaluation Criteria In Solid Tumors (RECIST version 1.1)
6. Expected survival >3 months
7. Women of child-bearing potential (i.e., women who are pre-menopausal or not surgically sterile) must use accepted highly effective contraceptive methods (abstinence, intrauterine device [IUD], oral contraceptive(s), intrauterine hormone releasing system (IUS), bilateral tubal occlusion or vasectomized partner) during and for 6 months after last study dose and must have a negative serum or urine pregnancy test within 1 week prior to treatment initiation, at monthly interval (day 1 of every even numbered cycle), at the end of systemic exposure, and at 30 days after the systemic exposure
8. Males with female partners (of childbearing potential) and female partners (of child bearing potential) with male partners must agree to use double barrier contraceptive measure (a combination of male condom with either cap, diaphragm or sponge with spermicide) in addition to oral contraception or avoidance of intercourse during the study and for 6 months after last study dose is received
9. At least 2 weeks must have elapsed from any prior surgery with resolution of any sequela for randomization
10. Laboratory values ≤2 weeks prior to randomization must be:

    * Adequate hematologic values

      * Platelet count ≥100,000 cells/mm3 or ≥100 bil/L;
      * Absolute neutrophil count [ANC] ≥1,500 cells/mm3 or ≥1.5 bil/L;
      * Hemoglobin ≥9 g/dL or ≥90 g/L)
    * Adequate hepatic function

      * Aspartate aminotransferase [AST/SGOT] ≤3x upper normal limit [UNL] (≤5x UNL if liver metastases present)
      * Alanine aminotransferase [ALT/SGPT] ≤3x UNL (≤5x UNL if liver metastases present)
      * Bilirubin (≤1.5x UNL); bilirubin ≤ 2.5 x ULN for subjects with Gilbert's syndrome
      * Serum albumin > 3.0 g/dL
    * Adequate renal function serum creatinine clearance CLcr > 30 mL/min). (Cocroft-Gault Formula should be used for CrCl calculation)
    * Adequate coagulation function • International Normalized Ratio or INR must be <1.5 unless on therapeutic blood thinners)
11. No evidence of active infection and no serious infection within the past 30 days.
12. Mentally competent, ability to understand and willingness to sign the informed consent form.

Exclusion Criteria:

1. Endocrine or acinar pancreatic carcinoma
2. Known cerebral metastases, central nervous system (CNS), or epidural tumor
3. Prior treatment with any chemotherapy for metastatic adenocarcinoma of the pancreas
4. Completion of a gemcitabine-based adjuvant chemotherapy regimen within less than 6 months at the time of screening.
5. Receipt of neoadjuvant or adjuvant FOLFIRINOX therapy if <6 months prior to disease recurrence
6. Patients with hypersensitivity to devimistat, FFX treatment or any of their excipients
7. Presence of clinically significant abdominal ascites
8. Patients receiving any other standard or investigational treatment for their cancer, or any other investigational agent for any indication within the past 2 weeks prior to initiation of devimistat treatment
9. Serious medical illness that would potentially increase patients' risk for toxicity
10. Any active uncontrolled bleeding, and any patients with a bleeding diathesis (e.g., active peptic ulcer disease)
11. Female patients who are pregnant or breastfeeding or planning to become pregnant or breastfeed during treatment and for an additional 6 months after the last dose of study treatment
12. Female patients of childbearing potential with a positive pregnancy test assessed by a serum pregnancy test at screening
13. Female patients of childbearing potential unwilling to use 1 highly effective method of contraception during treatment and for 6 months after the last dose of study treatment
14. Male patients with a pregnant partner who are unwilling to practice abstinence or use a condom during treatment and for 6 months after completion of study treatment
15. Male patients unwilling to abstain from donating sperm during treatment and for 6 months after completion of study treatment
16. Life expectancy less than 3 months
17. Any condition or abnormality which may, in the opinion of the investigator, compromise the safety of patients
18. Unwilling or unable to follow protocol requirements
19. Active heart disease including but not limited to symptomatic congestive heart failure (NYHA class 3 or 4), symptomatic coronary artery disease, symptomatic angina pectoris, or symptomatic myocardial infarction
20. Patients with a history of myocardial infarction that is <3 months prior to registration
21. Evidence of active infection, or serious infection within the past 30 days.
22. Patients with known HIV infection
23. Patients who have received cancer immunotherapy of any type within the past 2 weeks prior to initiation of devimistat treatment (steroids given for supportive care or in response to allergic reactions are allowed at any time)
24. Requirement for immediate palliative surgery, radiation or chemotherapy of any kind. Stenting for bile duct obstruction and need for pain medications are allowed provided all other inclusion criteria are met
25. Prior malignancy except for the following: adequately treated basal or squamous cell skin cancer, in situ cervical cancer, adequately treated cancer from which the patient has been disease-free for at least 3 years prior to screening
26. Unwilling or unable to avoid the concomitant use of strong CYP3A4 inducers or inhibitors during treatment with irinotecan
27. A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval > 480 milliseconds (ms) (CTCAE grade 1) using Fredericia's QT correction formula (i.e. QTcF)
28. A history of additional risk factors for TdP (e.g., heart failure, hypokalemia, family history of long QT syndrome)
29. The use of concomitant medications that prolong the QT/QTc intervals
30. Contraindications to any of the FFX treatment as follows:

Folinic Acid

* Calcium Folinate is contraindicated in patients who have previously shown hypersensitivity to folinate or any of the excipients.
* Calcium Folinate Injection is contraindicated in the treatment of pernicious anemia or other megaloblastic anemias where vitamin B12 is deficient. Its use can lead to an apparent response of the hematopoietic system, but neurological damage may occur or progress if already present.
* Patients with rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption should not take calcium folinate tablets.

Fluorouracil/5FU

* Fluorouracil is contraindicated in patients who have any known hypersensitivity to fluorouracil, are seriously debilitated or are suffering from bone marrow depression after radiotherapy or treatment with other antineoplastic agents, or who are suffering from a potentially serious infection.
* Fluorouracil is strictly contraindicated in pregnant or breast-feeding women.
* Flourouracil should not be used in the management of non-malignant disease.
* Fluorouracil must not be taken or used concomitantly with brivudin, sorivudine and analogues. Brivudin, sorivudine and analogues are potent inhibitors of the enzyme dihydropyrimidine dehydrogenase (DPD) which degrades fluorouracil
* In patients with known complete absence of dihydropyrimidine dehydrogenase (DPD) activity

Oxaliplatin

* Oxaliplatin is contraindicated in patients who have a known history of hypersensitivity to oxaliplatin or to any of the excipients
* are breast-feeding.
* have myelosuppression prior to starting first course, as evidenced by baseline neutrophils <2x109/l and/or platelet count of <100x109l.
* have a peripheral sensitive neuropathy with functional impairment prior to first course.
* have a severely impaired renal function (creatinine clearance less than 30 ml /min)

Irinotecan

* Chronic inflammatory bowel disease and/or bowel obstruction
* History of severe hypersensitivity reactions to Irinotecan hydrochloride trihydrate or to any of the excipients
* Bilirubin > 3 times the ULN
* Severe bone marrow failure.
* WHO performance status > 2.
* Concomitant use with St John's wort

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 528 (Actual)
Dates: Start 2018-11-09 (Actual); Primary Completion 2021-08-16 (Actual); Study Completion 2022-01-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip A Philip, MD, PhD, FRCP, Principal Investigator — Karmanos Cancer Institute at Wayne State University
Locations (74):
- United States (40):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - The University of Arizona Cancer Center, Tucson, Arizona
  - City of Hope, Duarte, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - UCLA Medical Center, Los Angeles, California
  - Pacific Hematology Oncology Associates, San Francisco, California
  - Smilow Cancer Hospital at Yale-New Haven, New Haven, Connecticut
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Mayo Clinic Hospital, Jacksonville, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Northwestern Memorial Hospital - Arkes Family Pavilion, Chicago, Illinois
  - University of Chicago, Harvey, Illinois
  - The University of Kansas Cancer Center - Clinical Research Center - Fairway Office Park, Fairway, Kansas
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - University of Micihgan, Ann Arbor, Michigan
  - Karmanos cancer Center, Detroit, Michigan
  - Mayo Clinic Cancer Center (MCCC), Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Comprehensive Cancer centers of Nevada, Las Vegas, Nevada
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - Atlantic Health System, Morristown, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - New York University Langone Medical Center, New York, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Levine cancer Institute, Charlotte, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - University of Cincinnati Cancer Institute, Cincinnati, Ohio
  - Cleveland Clinic - Taussig Cancer Center, Cleveland, Ohio
  - University Hospitals - Seidman Cancer Center, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - University of Pittsburgh-Hillman cancer ceter, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center-Vanderbilt-Ingram Cancer Center-Henry-Joyce Cancer Clinic, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Huntsman cancer Institute, Salt Lake City, Utah
  - University of Virginia Cancer Center - Emily Couric Clinical Cancer Center, Charlottesville, Virginia
  - VCU Massey Cancer Center, Richmond, Virginia
  - Blue Ridge Cancer Care, Roanoke, Virginia
  - Seattle Cancer Care Alliance, Seattle, Washington
- Belgium (2):
  - Hôpital Erasme, Brussels, Brussels Capital
  - UZ Leuven, Leuven, VBR
- France (10):
  - CHRU Brest - Hôpital Morvan, Brest
  - Hôpital Beaujon, Clichy
  - Centre Hospitalier Départemental Vendée - Hôpital de la Roche-sur-Yon, La Roche-sur-Yon
  - L'ICM, Institut régional du Cancer de Montpellier, Montpellier
  - CHU de Nantes - Hôpital Nord Laennec, Nantes
  - CHU Hopitaux de Bordeaux - Hôpital Saint-André, Pessac
  - CHU de Poitiers, Poitiers
  - Centre Eugène Marquis, Rennes
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - Gustave Roussy Cancer Campus Grand Paris (Institut de Cancerologie Gustave-Roussy), Villejuif
- Germany (3):
  - SLK-Kliniken Heilbronn GmbH, Heilbronn, Baden-Wurttemberg
  - Universitätsklinikum Knappschaftskrankenhaus Bochum GmbH, Bochum
  - Universitaetsklinikum Tuebingen, Tübingen
- Israel (7):
  - Hillel Yaffe Medical Center, Hadera, Haifa District
  - Rambam Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Sanz Medical Center - Laniado Hospital, Netanya
  - The Chaim Sheba Medical Center - Sheba Cancer Research Center (SCRC), Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - Assaf-Harofeh Medical Center, Ẕerifin
- South Korea (12):
  - The Catholic University of Korea - Seoul St. Mary's Hospital (Kangnam St. Mary's Hospital), Seocho, Seoul
  - Seoul National University Hospital, Busan
  - Kyungpook National University Chilgok Hospital, Daegu
  - Gachon University Gil Hospital, Incheon
  - Inha University Hospital, Incheon
  - Seoul National University Bundang Hospital, Seongnam-si
  - Seoul National University Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Severance Hospital - Yonsei Cancer Center, Seoul
  - Samsung Medical Center, Seoul
  - National Cancer Center, Seoul
  - Ajou University Hospital, Suwon

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Philip PA, Sahai V, Bahary N, Mahipal A, Kasi A, Rocha Lima CMS, Alistar AT, Oberstein PE, Golan T, Metges JP, Lacy J, Fountzilas C, Lopez CD, Ducreux M, Hammel P, Salem M, Bajor D, Benson AB, Luther S, Pardee T, Van Cutsem E. Devimistat (CPI-613) With Modified Fluorouarcil, Oxaliplatin, Irinotecan, and Leucovorin (FFX) Versus FFX for Patients With Metastatic Adenocarcinoma of the Pancreas: The Phase III AVENGER 500 Study. J Clin Oncol. 2024 Nov;42(31):3692-3701. doi: 10.1200/JCO.23.02659. Epub 2024 Aug 1. PMID 39088774
- [Derived] Liu N, Yan M, Tao Q, Wu J, Chen J, Chen X, Peng C. Inhibition of TCA cycle improves the anti-PD-1 immunotherapy efficacy in melanoma cells via ATF3-mediated PD-L1 expression and glycolysis. J Immunother Cancer. 2023 Sep;11(9):e007146. doi: 10.1136/jitc-2023-007146. PMID 37678921
- [Derived] Philip PA, Buyse ME, Alistar AT, Rocha Lima CM, Luther S, Pardee TS, Van Cutsem E. A Phase III open-label trial to evaluate efficacy and safety of CPI-613 plus modified FOLFIRINOX (mFFX) versus FOLFIRINOX (FFX) in patients with metastatic adenocarcinoma of the pancreas. Future Oncol. 2019 Oct;15(28):3189-3196. doi: 10.2217/fon-2019-0209. Epub 2019 Sep 12. PMID 31512497

RESULTS

PARTICIPANT FLOW:
Groups:
- CPI-613, mFolfirinox: CPI-613, mFolfirinox
  CPI-613 at 500 mg/m2 IV infusion at a rate of 4mL/min via a central venous port on day 1 and 3 of a 14-day cycle.
  mFolfirinox (given immediately after CPI-613 administration): Oxaliplatin (Eloxatin) at 65 mg/m2 given as a 2 hr IV infusion, Folinic acid at 400 mg/m2 given as a 90 min (1.5hr) infusion immediately after Oxaliplatin, and concurrently with Irinotecan (irinotecan at 140mg/m2 given as a 90 min IV infusion) via a Y-connector, Flurouracil at 400 mg/m2 as bolus followed by a 46 hr infusion at 2400mg/m2 starting immediately after completion of folinic acid and Irinotecan.
  CPI 613, mFolfirinox: CPI-613: 500mg/m2, IV infusion at a rate of 4mL/min via a central venous port.
  mFolfirinox: given immediately after CPI-613 administration
- Folfirinox: Folfirinox
  Folfirinox: Oxaliplatin (Eloxatin) at 85 mg/m2 given as a 2 hr IV infusion, Folinic acid at 400 mg/m2 given as a 90 min (1.5hr) infusion immediately after Oxaliplatin, and concurrently with Irinotecan (irinotecan at 180mg/m2 given as a 90 min IV infusion) via a Y-connector, Flurouracil at 400 mg/m2 as bolus followed by a 46 hr infusion at 2400mg/m2 starting immediately after completion of folinic acid and Irinotecan.
  Folfirinox: Folfirinox
Period: Overall Study
Arm/Group | CPI-613, mFolfirinox | Folfirinox
Started | 266 | 262
Completed | 259 | 235
Not Completed | 7 | 27

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CPI-613, mFolfirinox | Folfirinox | Total
Number analyzed (Participants) | 266 | 262 | 528
Age, Customized [Mean (Standard Deviation); unit: years] | 61.62 (8.67) | 61.47 (8.30) | 61.55 (8.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 112 | 102 | 214
  Male | 154 | 160 | 314
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 31 | 30 | 61
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 10 | 7 | 17
  White | 201 | 200 | 401
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 23 | 24 | 47

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Defined as the duration from the date of randomization to the date of death from any cause
Time Frame: 38 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | CPI-613, mFolfirinox | Folfirinox
Number analyzed (Participants) | 266 | 262
months | 11.10 [10.22 to 12.94] | 11.73 [10.12 to 13.24]

2. Secondary Outcome: Progression Free Survival (PFS)
Description: Defined as the duration from the date of randomization to the date of progressive disease or death from any cause.
  Progressive Disease is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as at least 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must have also demonstrated an absolute increase of at least 5 mm. The appearance of one or more new lesions was also considered progression.
Time Frame: 38 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | CPI-613, mFolfirinox | Folfirinox
Number analyzed (Participants) | 266 | 262
months | 7.82 [6.97 to 10.91] | 7.98 [7.23 to 11.14]

3. Secondary Outcome: Overall Response Rate (ORR)
Description: Defined as the rate of Complete Response (CR) plus Partial Response (PR): Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), at least 30% decrease in the sum of diameters of target lesions;
Time Frame: 38 months
Measure: Count of Participants; unit: Participants
Arm/Group | CPI-613, mFolfirinox | Folfirinox
Number analyzed (Participants) | 266 | 262
Participants | 104 | 90

ADVERSE EVENTS:
Time Frame: 38 months
Arm/Group | CPI-613, mFolfirinox | Folfirinox
All-Cause Mortality (participants affected / at risk) | 140/259 | 133/235
Serious Adverse Events (participants affected / at risk) | 140/259 | 133/235
Other Adverse Events (participants affected / at risk) | 258/259 | 232/235
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CPI-613, mFolfirinox (N=259) | Folfirinox (N=235)
Anaemia (Blood and lymphatic system disorders) | 10 | 21
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 3
Leukocytosis (Blood and lymphatic system disorders) | 3 | 17
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 2 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 3
Acute left ventricular failure (Cardiac disorders) | 2 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Arteriospasm coronary (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Atrial flutter (Cardiac disorders) | 1 | 3
Atrial thrombosis (Cardiac disorders) | 1 | 1
Atrioventricular block complete (Cardiac disorders) | 1 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0
Stress cardiomyopathy (Cardiac disorders) | 2 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Meniere's disease (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 15 | 10
Ascites (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 5 | 5
Constipation (Gastrointestinal disorders) | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 9 | 18
Duodenal obstruction (Gastrointestinal disorders) | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 2 | 0
Enterocolitis (Gastrointestinal disorders) | 3 | 1
Gastric varices haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastroduodenal ulcer (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 | 4
Haematochezia (Gastrointestinal disorders) | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 2 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Large intestine perforation (Gastrointestinal disorders) | 2 | 0
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 7 | 6
Obstruction gastric (Gastrointestinal disorders) | 1 | 2
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 1
Pancreatic duct dilatation (Gastrointestinal disorders) | 1 | 0
Pancreatic necrosis (Gastrointestinal disorders) | 1 | 0
Pancreatic pseudocyst (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 2 | 2
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 6
Subileus (Gastrointestinal disorders) | 1 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 | 0
Vomiting (Gastrointestinal disorders) | 7 | 8
Asthenia (General disorders) | 0 | 3
Device related thrombosis (General disorders) | 0 | 1
Drug intolerance (General disorders) | 1 | 1
Fatigue (General disorders) | 1 | 1
General physical health deterioration (General disorders) | 5 | 4
Hyperthermia (General disorders) | 0 | 1
Incarcerated hernia (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 4
Sudden death (General disorders) | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 0 | 1
Vascular stent stenosis (General disorders) | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 5 | 4
Bile duct stenosis (Hepatobiliary disorders) | 0 | 1
Biliary dilatation (Hepatobiliary disorders) | 1 | 0
Biliary tract disorder (Hepatobiliary disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 8
Cholangitis acute (Hepatobiliary disorders) | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 5 | 3
Cholestasis (Hepatobiliary disorders) | 0 | 1
Gallbladder obstruction (Hepatobiliary disorders) | 2 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 2
Jaundice (Hepatobiliary disorders) | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 1
Liver injury (Hepatobiliary disorders) | 0 | 1
Malignant biliary obstruction (Hepatobiliary disorders) | 1 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 1
Abdominal infection (Infections and infestations) | 0 | 1
Arthritis bacterial (Infections and infestations) | 1 | 0
Arthritis infective (Infections and infestations) | 1 | 1
Bacteraemia (Infections and infestations) | 4 | 2
Biliary tract infection (Infections and infestations) | 2 | 1
Cholecystitis infective (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Corona virus infection (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 4 | 0
Endocarditis (Infections and infestations) | 1 | 0
Enteritis infectious (Infections and infestations) | 0 | 1
Enterocolitis infectious (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 0 | 1
Fungal infection (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 3
H1N1 influenza (Infections and infestations) | 0 | 1
Infected skin ulcer (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 2 | 0
Klebsiella bacteraemia (Infections and infestations) | 1 | 0
Liver abscess (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 0 | 1
Neutropenic sepsis (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 0 | 1
Peritonitis bacterial (Infections and infestations) | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 3 | 6
Pneumonia viral (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 10 | 4
Septic shock (Infections and infestations) | 6 | 2
Subcutaneous abscess (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 2
Urosepsis (Infections and infestations) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Shunt malfunction (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 3
Blood creatinine increased (Investigations) | 2 | 0
Blood glucose increased (Investigations) | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 2 | 3
Platelet count decreased (Investigations) | 2 | 3
Transaminases increased (Investigations) | 0 | 1
Weight decreased (Investigations) | 1 | 0
White blood cell count decreased (Investigations) | 1 | 2
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 4 | 3
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 | 1
Failure to thrive (Metabolism and nutrition disorders) | 1 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0
Hypophagia (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Chest wall haematoma (Musculoskeletal and connective tissue disorders) | 0 | 1
Fistula (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 3 | 1
Encephalopathy (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 3 | 0
Device occlusion (Product Issues) | 1 | 2
Stent malfunction (Product Issues) | 1 | 1
Confusional state (Psychiatric disorders) | 1 | 1
Delirium (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 2 | 0
Mental status changes (Psychiatric disorders) | 2 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Embolism (Vascular disorders) | 2 | 1
Hypertension (Vascular disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 10 | 1
Hypotension (Vascular disorders) | 1 | 2
Vena cava thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CPI-613, mFolfirinox (N=259) | Folfirinox (N=235)
Anaemia (Blood and lymphatic system disorders) | 120 | 94
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 7 | 19
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 8 | 7
Leukopenia (Blood and lymphatic system disorders) | 2 | 1
Lymph node pain (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 3 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 48 | 49
Normocytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 2 | 4
Splenic infarction (Blood and lymphatic system disorders) | 1 | 1
Splenic vein thrombosis (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 34 | 38
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 0
Acute left ventricular failure (Cardiac disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 1
Arteriospasm coronary (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 6 | 7
Atrial flutter (Cardiac disorders) | 1 | 1
Atrial thrombosis (Cardiac disorders) | 1 | 1
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 6 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac disorder (Cardiac disorders) | 1 | 0
Cardiac ventricular thrombosis (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Coronary artery thrombosis (Cardiac disorders) | 1 | 0
Intracardiac mass (Cardiac disorders) | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 1
Left ventricular failure (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 6 | 2
Sinus bradycardia (Cardiac disorders) | 5 | 3
Sinus tachycardia (Cardiac disorders) | 12 | 8
Stress cardiomyopathy (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 8 | 4
Ventricular extrasystoles (Cardiac disorders) | 2 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Congenital, familial and genetic disorders (Cardiac disorders) | 1 | 0
Hereditary non-polyposis colorectal cancer syndrome (Cardiac disorders) | 1 | 0
Dacryostenosis acquired (Ear and labyrinth disorders) | 0 | 1
Dry eye (Ear and labyrinth disorders) | 3 | 6
Dyschromatopsia (Ear and labyrinth disorders) | 1 | 0
Eye pain (Ear and labyrinth disorders) | 2 | 0
Eye swelling (Ear and labyrinth disorders) | 1 | 0
Glaucoma (Ear and labyrinth disorders) | 1 | 0
Lacrimation increased (Ear and labyrinth disorders) | 2 | 0
Ocular hyperaemia (Ear and labyrinth disorders) | 2 | 0
Periorbital oedema (Ear and labyrinth disorders) | 1 | 0
Photophobia (Ear and labyrinth disorders) | 2 | 0
Retinal detachment (Ear and labyrinth disorders) | 1 | 0
Swelling of eyelid (Ear and labyrinth disorders) | 1 | 0
Vision blurred (Ear and labyrinth disorders) | 11 | 4
Visual acuity reduced (Ear and labyrinth disorders) | 1 | 0
Visual impairment (Ear and labyrinth disorders) | 5 | 2
Vitreous floaters (Ear and labyrinth disorders) | 1 | 2
Xerophthalmia (Ear and labyrinth disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 7 | 5
Abdominal distension (Gastrointestinal disorders) | 25 | 17
Abdominal hernia (Gastrointestinal disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 90 | 84
Abdominal pain lower (Gastrointestinal disorders) | 5 | 4
Abdominal pain upper (Gastrointestinal disorders) | 22 | 11
Abdominal rigidity (Gastrointestinal disorders) | 1 | 5
Abdominal tenderness (Gastrointestinal disorders) | 1 | 0
Abnormal faeces (Gastrointestinal disorders) | 2 | 1
Anal fissure (Gastrointestinal disorders) | 1 | 4
Anal haemorrhage (Gastrointestinal disorders) | 1 | 2
Anal incontinence (Gastrointestinal disorders) | 1 | 2
Anal ulcer (Gastrointestinal disorders) | 0 | 1
Aphthous ulcer (Gastrointestinal disorders) | 2 | 0
Ascites (Gastrointestinal disorders) | 15 | 11
Bowel movement irregularity (Gastrointestinal disorders) | 1 | 1
Chapped lips (Gastrointestinal disorders) | 0 | 1
Cheilitis (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 8 | 5
Constipation (Gastrointestinal disorders) | 95 | 67
Diarrhoea (Gastrointestinal disorders) | 174 | 174
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 19 | 12
Dumping syndrome (Gastrointestinal disorders) | 0 | 1
Duodenal obstruction (Gastrointestinal disorders) | 2 | 2
Dyspepsia (Gastrointestinal disorders) | 30 | 25
Dysphagia (Gastrointestinal disorders) | 11 | 10
Enteritis (Gastrointestinal disorders) | 3 | 0
Enterocolitis (Gastrointestinal disorders) | 3 | 1
Epigastric discomfort (Gastrointestinal disorders) | 1 | 1
Eructation (Gastrointestinal disorders) | 4 | 3
Faeces discoloured (Gastrointestinal disorders) | 1 | 1
Faeces pale (Gastrointestinal disorders) | 3 | 0
Flatulence (Gastrointestinal disorders) | 21 | 14
Frequent bowel movements (Gastrointestinal disorders) | 1 | 1
Gastric polyps (Gastrointestinal disorders) | 0 | 1
Gastric varices (Gastrointestinal disorders) | 0 | 2
Gastric varices haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 5 | 1
Gastritis erosive (Gastrointestinal disorders) | 0 | 1
Gastroduodenal ulcer (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 | 4
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 | 2
Gastrointestinal pain (Gastrointestinal disorders) | 2 | 2
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 24 | 21
Gingival bleeding (Gastrointestinal disorders) | 0 | 2
Gingival pain (Gastrointestinal disorders) | 2 | 1
Gingival recession (Gastrointestinal disorders) | 1 | 0
Glossitis (Gastrointestinal disorders) | 1 | 0
Glossodynia (Gastrointestinal disorders) | 2 | 0
Haematemesis (Gastrointestinal disorders) | 2 | 2
Haematochezia (Gastrointestinal disorders) | 10 | 3
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 2 | 2
Haemorrhoids (Gastrointestinal disorders) | 11 | 13
Hypoaesthesia oral (Gastrointestinal disorders) | 1 | 2
Ileus (Gastrointestinal disorders) | 1 | 2
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 3 | 1
Intra-abdominal fluid collection (Gastrointestinal disorders) | 0 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Large intestine perforation (Gastrointestinal disorders) | 2 | 0
Lip dry (Gastrointestinal disorders) | 1 | 0
Lip oedema (Gastrointestinal disorders) | 1 | 1
Lip swelling (Gastrointestinal disorders) | 1 | 1
Lip ulceration (Gastrointestinal disorders) | 2 | 3
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 3 | 1
Mesenteric vein thrombosis (Gastrointestinal disorders) | 1 | 1
Mouth ulceration (Gastrointestinal disorders) | 3 | 0
Nausea (Gastrointestinal disorders) | 193 | 155
Obstruction gastric (Gastrointestinal disorders) | 2 | 2
Odynophagia (Gastrointestinal disorders) | 2 | 0
Oesophageal achalasia (Gastrointestinal disorders) | 0 | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 4 | 3
Oral dysaesthesia (Gastrointestinal disorders) | 1 | 2
Oral mucosal eruption (Gastrointestinal disorders) | 1 | 0
Oral pain (Gastrointestinal disorders) | 9 | 4
Pancreatic duct dilatation (Gastrointestinal disorders) | 1 | 0
Pancreatic failure (Gastrointestinal disorders) | 2 | 4
Pancreatic necrosis (Gastrointestinal disorders) | 1 | 0
Pancreatic pseudocyst (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 2 | 2
Paraesthesia oral (Gastrointestinal disorders) | 4 | 1
Periodontal disease (Gastrointestinal disorders) | 0 | 2
Pneumatosis intestinalis (Gastrointestinal disorders) | 1 | 0
Proctalgia (Gastrointestinal disorders) | 6 | 5
Rectal haemorrhage (Gastrointestinal disorders) | 4 | 3
Reflux gastritis (Gastrointestinal disorders) | 1 | 0
Retching (Gastrointestinal disorders) | 0 | 2
Saliva altered (Gastrointestinal disorders) | 0 | 1
Salivary hypersecretion (Gastrointestinal disorders) | 3 | 4
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 7
Steatorrhoea (Gastrointestinal disorders) | 2 | 2
Stomatitis (Gastrointestinal disorders) | 52 | 47
Subileus (Gastrointestinal disorders) | 1 | 1
Swollen tongue (Gastrointestinal disorders) | 1 | 1
Tongue discolouration (Gastrointestinal disorders) | 1 | 1
Tongue disorder (Gastrointestinal disorders) | 0 | 1
Tongue dry (Gastrointestinal disorders) | 1 | 0
Tongue oedema (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 2 | 4
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 | 0
Vomiting (Gastrointestinal disorders) | 107 | 96
Administration site extravasation (General disorders) | 1 | 0
Asthenia (General disorders) | 34 | 46
Catheter site discolouration (General disorders) | 0 | 1
Catheter site erythema (General disorders) | 0 | 1
Catheter site inflammation (General disorders) | 1 | 0
Catheter site oedema (General disorders) | 1 | 0
Catheter site pain (General disorders) | 4 | 2
Catheter site thrombosis (General disorders) | 0 | 1
Chest discomfort (General disorders) | 3 | 2
Chest pain (General disorders) | 1 | 0
Chills (General disorders) | 16 | 13
Complication associated with device (General disorders) | 1 | 0
Device embolisation (General disorders) | 0 | 1
Device related thrombosis (General disorders) | 2 | 2
Discomfort (General disorders) | 1 | 0
Drug intolerance (General disorders) | 1 | 1
Early satiety (General disorders) | 3 | 4
Facial pain (General disorders) | 1 | 0
Fatigue (General disorders) | 153 | 126
Feeling cold (General disorders) | 2 | 2
Feeling hot (General disorders) | 1 | 2
Gait disturbance (General disorders) | 3 | 0
General physical health deterioration (General disorders) | 7 | 4
Generalised oedema (General disorders) | 2 | 2
Hernia (General disorders) | 0 | 1
Hyperthermia (General disorders) | 0 | 1
Incarcerated hernia (General disorders) | 1 | 0
Influenza like illness (General disorders) | 1 | 3
Injection site reaction (General disorders) | 1 | 1
Localised oedema (General disorders) | 6 | 3
Malaise (General disorders) | 3 | 8
Mucosal inflammation (General disorders) | 26 | 22
Non-cardiac chest pain (General disorders) | 15 | 7
Oedema (General disorders) | 3 | 4
Oedema peripheral (General disorders) | 44 | 36
Pain (General disorders) | 6 | 7
Performance status decreased (General disorders) | 0 | 1
Peripheral swelling (General disorders) | 4 | 2
Pyrexia (General disorders) | 40 | 41
Sensation of foreign body (General disorders) | 1 | 0
Sudden death (General disorders) | 1 | 0
Swelling (General disorders) | 3 | 0
Systemic inflammatory response syndrome (General disorders) | 1 | 1
Temperature intolerance (General disorders) | 31 | 21
Unevaluable event (General disorders) | 1 | 0
Vascular stent stenosis (General disorders) | 0 | 1
Xerosis (General disorders) | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 6 | 5
Bile duct stenosis (Hepatobiliary disorders) | 1 | 1
Biliary dilatation (Hepatobiliary disorders) | 2 | 0
Biliary tract disorder (Hepatobiliary disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 2 | 11
Cholangitis acute (Hepatobiliary disorders) | 2 | 1
Cholecystitis (Hepatobiliary disorders) | 6 | 3
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Cholestasis (Hepatobiliary disorders) | 4 | 2
Gallbladder obstruction (Hepatobiliary disorders) | 2 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Hepatic pain (Hepatobiliary disorders) | 1 | 0
Hepatic steatosis (Hepatobiliary disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0
Hepatocellular injury (Hepatobiliary disorders) | 2 | 5
Hyperbilirubinaemia (Hepatobiliary disorders) | 7 | 3
Ischaemic hepatitis (Hepatobiliary disorders) | 2 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 2 | 1
Liver injury (Hepatobiliary disorders) | 0 | 1
Malignant biliary obstruction (Hepatobiliary disorders) | 1 | 0
Ocular icterus (Hepatobiliary disorders) | 1 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 4
Immune system disorders (Hepatobiliary disorders) | 5 | 9
Anaphylactic reaction (Hepatobiliary disorders) | 0 | 1
Drug hypersensitivity (Hepatobiliary disorders) | 2 | 3
Hypersensitivity (Hepatobiliary disorders) | 3 | 3
Seasonal allergy (Hepatobiliary disorders) | 0 | 3
Abdominal infection (Infections and infestations) | 0 | 2
Abscess (Infections and infestations) | 2 | 0
Angular cheilitis (Infections and infestations) | 0 | 1
Arthritis bacterial (Infections and infestations) | 1 | 0
Arthritis infective (Infections and infestations) | 1 | 1
Asymptomatic bacteriuria (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 6 | 3
Bacterial colitis (Infections and infestations) | 1 | 0
Bacterial infection (Infections and infestations) | 1 | 0
Biliary tract infection (Infections and infestations) | 2 | 1
Bronchiolitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Candida infection (Infections and infestations) | 7 | 2
Catheter site infection (Infections and infestations) | 4 | 0
Cellulitis (Infections and infestations) | 3 | 1
Cholecystitis infective (Infections and infestations) | 1 | 0
Clostridial infection (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 2 | 1
Clostridium difficile infection (Infections and infestations) | 3 | 0
Conjunctivitis (Infections and infestations) | 1 | 0
Corona virus infection (Infections and infestations) | 6 | 2
Cytomegalovirus colitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 4 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Ear infection (Infections and infestations) | 1 | 1
Endocarditis (Infections and infestations) | 1 | 0
Enteritis infectious (Infections and infestations) | 0 | 1
Enterocolitis infectious (Infections and infestations) | 1 | 0
Enterovirus infection (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 0 | 2
Escherichia bacteraemia (Infections and infestations) | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 1 | 0
Folliculitis (Infections and infestations) | 1 | 0
Fungal infection (Infections and infestations) | 1 | 1
Fungal oesophagitis (Infections and infestations) | 1 | 0
Fungal skin infection (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 2 | 3
Gingival abscess (Infections and infestations) | 1 | 0
Gingivitis (Infections and infestations) | 1 | 0
H1N1 influenza (Infections and infestations) | 0 | 1
Herpes simplex (Infections and infestations) | 3 | 0
Herpes virus infection (Infections and infestations) | 1 | 1
Herpes zoster (Infections and infestations) | 2 | 3
Hordeolum (Infections and infestations) | 0 | 2
Infected cyst (Infections and infestations) | 1 | 0
Infected skin ulcer (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 1
Influenza (Infections and infestations) | 4 | 1
Klebsiella bacteraemia (Infections and infestations) | 1 | 0
Liver abscess (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 4
Mucosal infection (Infections and infestations) | 1 | 1
Myelitis (Infections and infestations) | 1 | 0
Nail infection (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 4
Neutropenic sepsis (Infections and infestations) | 1 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 2
Oral candidiasis (Infections and infestations) | 5 | 8
Oral fungal infection (Infections and infestations) | 4 | 3
Oral herpes (Infections and infestations) | 4 | 1
Oropharyngeal candidiasis (Infections and infestations) | 1 | 0
Paronychia (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 0 | 1
Peritonitis bacterial (Infections and infestations) | 1 | 2
Pharyngitis (Infections and infestations) | 2 | 0
Pharyngitis streptococcal (Infections and infestations) | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 8 | 12
Pneumonia viral (Infections and infestations) | 0 | 1
Rash pustular (Infections and infestations) | 3 | 0
Rhinitis (Infections and infestations) | 7 | 2
Rhinovirus infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 11 | 6
Septic shock (Infections and infestations) | 6 | 2
Sinusitis (Infections and infestations) | 3 | 1
Skin infection (Infections and infestations) | 1 | 1
Subcutaneous abscess (Infections and infestations) | 1 | 2
Tinea pedis (Infections and infestations) | 0 | 2
Tongue fungal infection (Infections and infestations) | 0 | 2
Tonsillitis (Infections and infestations) | 0 | 2
Tooth abscess (Infections and infestations) | 1 | 0
Tooth infection (Infections and infestations) | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 8 | 5
Urinary tract infection (Infections and infestations) | 9 | 12
Urosepsis (Infections and infestations) | 0 | 1
Vaginal infection (Infections and infestations) | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 2 | 4
Vulvovaginitis (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 1 | 0
Abdominal injury (Injury, poisoning and procedural complications) | 0 | 1
Animal bite (Injury, poisoning and procedural complications) | 1 | 0
Burn oesophageal (Injury, poisoning and procedural complications) | 1 | 0
Compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 7 | 4
Fall (Injury, poisoning and procedural complications) | 12 | 4
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Foreign body in respiratory tract (Injury, poisoning and procedural complications) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 1
Gingival injury (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 16 | 22
Ligament sprain (Injury, poisoning and procedural complications) | 2 | 0
Limb injury (Injury, poisoning and procedural complications) | 2 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Post procedural bile leak (Injury, poisoning and procedural complications) | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 2 | 0
Procedural dizziness (Injury, poisoning and procedural complications) | 0 | 1
Procedural hypertension (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 2 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Seroma (Injury, poisoning and procedural complications) | 1 | 0
Shunt malfunction (Injury, poisoning and procedural complications) | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Sunburn (Injury, poisoning and procedural complications) | 0 | 1
Testicular injury (Injury, poisoning and procedural complications) | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 3 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 3 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1
Transfusion related complication (Injury, poisoning and procedural complications) | 0 | 1
Urethral injury (Injury, poisoning and procedural complications) | 1 | 0
Vaccination complication (Injury, poisoning and procedural complications) | 1 | 1
Vascular access complication (Injury, poisoning and procedural complications) | 1 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 1
Activated partial thromboplastin time prolonged (Investigations) | 24 | 15
Alanine aminotransferase increased (Investigations) | 60 | 41
Amylase increased (Investigations) | 1 | 1
Anion gap decreased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 57 | 33
Bacterial test positive (Investigations) | 0 | 1
Band neutrophil percentage increased (Investigations) | 1 | 0
Blood albumin decreased (Investigations) | 3 | 1
Blood alkaline phosphatase increased (Investigations) | 71 | 44
Blood bilirubin decreased (Investigations) | 2 | 0
Blood bilirubin increased (Investigations) | 15 | 17
blood calcium decreased (Investigations) | 1 | 0
blood chloride decreased (Investigations) | 1 | 0
blood chloride increased (Investigations) | 1 | 0
blood cholesterol increased (Investigations) | 2 | 1
blood creatinine decreased (Investigations) | 1 | 1
blood creatinine increased (Investigations) | 10 | 15
blood fibrinogen decreased (Investigations) | 0 | 1
blood glucose increased (Investigations) | 0 | 3
blood iron decreased (Investigations) | 1 | 0
blood lactic acid increased (Investigations) | 0 | 1
blood magnesium decreased (Investigations) | 2 | 0
blood phosphorus decreased (Investigations) | 4 | 1
blood phosphorus increased (Investigations) | 0 | 2
blood potassium decreased (Investigations) | 1 | 2
bloo pressure increased (Investigations) | 0 | 1
Blood pressure orthostatic decreased (Investigations) | 0 | 1
Blood sodium decreased (Investigations) | 2 | 2
Blood urea decreased (Investigations) | 1 | 0
Blood urea increased (Investigations) | 0 | 1
C-reactive protein increased (Investigations) | 0 | 1
Cardiac murmur (Investigations) | 2 | 1
Catheterisation cardiac (Investigations) | 0 | 1
Coronavirus test positive (Investigations) | 1 | 0
Ejection fraction decreased (Investigations) | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 4 | 1
Electrocardiogram T wave inversion (Investigations) | 0 | 1
Fibrin D dimer increased (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 4 | 2
Grip strength decreased (Investigations) | 0 | 1
Haematocrit decreased (Investigations) | 0 | 1
Heart rate increased (Investigations) | 3 | 1
Hepatic enzyme increased (Investigations) | 2 | 2
Immature granulocyte count increased (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 24 | 25
Lipase increased (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 37 | 23
Lymphocyte count increased (Investigations) | 4 | 1
Mean cell volume increased (Investigations) | 1 | 0
Metamyelocyte count increased (Investigations) | 1 | 0
Monocyte count decreased (Investigations) | 1 | 0
Monocyte count increased (Investigations) | 1 | 1
Neutrophil count decreased (Investigations) | 73 | 61
Neutrophil count increased (Investigations) | 4 | 2
Pancreatic enzymes decreased (Investigations) | 4 | 5
Platelet count decreased (Investigations) | 80 | 67
Platelet count increased (Investigations) | 1 | 0
Prostatic specific antigen increased (Investigations) | 1 | 0
Protein total decreased (Investigations) | 2 | 4
Prothrombin time prolonged (Investigations) | 2 | 1
Red blood cell count decreased (Investigations) | 0 | 1
Red blood cell count increased (Investigations) | 0 | 1
Transaminases increased (Investigations) | 2 | 3
Troponin increased (Investigations) | 0 | 1
Urine output decreased (Investigations) | 1 | 1
Weight decreased (Investigations) | 87 | 78
Weight increased (Investigations) | 11 | 4
White blood cell count decreased (Investigations) | 40 | 34
White blood cell count increased (Investigations) | 4 | 1
Abnormal loss of weight (Metabolism and nutrition disorders) | 1 | 0
Acidosis (Metabolism and nutrition disorders) | 1 | 1
Cachexia (Metabolism and nutrition disorders) | 1 | 0
Cell death (Metabolism and nutrition disorders) | 1 | 2
Decreased appetite (Metabolism and nutrition disorders) | 111 | 102
Dehydration (Metabolism and nutrition disorders) | 38 | 36
Diabetes mellitus (Metabolism and nutrition disorders) | 7 | 4
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 2
Food intolerance (Metabolism and nutrition disorders) | 0 | 1
Glucose tolerance impaired (Metabolism and nutrition disorders) | 2 | 1
Gout (Metabolism and nutrition disorders) | 2 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 3 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 33 | 24
Hyperkalaemia (Metabolism and nutrition disorders) | 11 | 10
Hypermagnesaemia (Metabolism and nutrition disorders) | 6 | 5
Hypernatraemia (Metabolism and nutrition disorders) | 7 | 4
Hyperphosphataemia (Metabolism and nutrition disorders) | 5 | 3
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 54 | 42
Hypocalcaemia (Metabolism and nutrition disorders) | 32 | 24
Hypoglycaemia (Metabolism and nutrition disorders) | 11 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 96 | 87
Hypomagnesaemia (Metabolism and nutrition disorders) | 46 | 49
Hyponatraemia (Metabolism and nutrition disorders) | 52 | 39
Hypophagia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 41 | 30
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 1
Iron deficiency (Metabolism and nutrition disorders) | 0 | 2
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 5 | 4
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0
Pseudohyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 1
Vitamin K deficiency (Metabolism and nutrition disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 18 | 14
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 43 | 36
Bone pain (Musculoskeletal and connective tissue disorders) | 5 | 5
Chest wall haematoma (Musculoskeletal and connective tissue disorders) | 0 | 1
Fistula (Musculoskeletal and connective tissue disorders) | 2 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 9 | 5
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 | 2
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 2
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 11 | 11
Muscle twitching (Musculoskeletal and connective tissue disorders) | 3 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 16 | 12
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 5 | 4
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 8 | 10
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 16 | 8
Neck pain (Musculoskeletal and connective tissue disorders) | 6 | 6
Osteitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 | 8
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 10
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1 | 1
Benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Haemangioma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Ageusia (Nervous system disorders) | 0 | 1
Amnesia (Nervous system disorders) | 1 | 0
Aphasia (Nervous system disorders) | 2 | 2
Ataxia (Nervous system disorders) | 2 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 3 | 2
Cholinergic syndrome (Nervous system disorders) | 12 | 11
Cognitive disorder (Nervous system disorders) | 1 | 1
Disturbance in attention (Nervous system disorders) | 4 | 1
Dizziness (Nervous system disorders) | 50 | 32
Dizziness postural (Nervous system disorders) | 2 | 0
Dysaesthesia (Nervous system disorders) | 5 | 12
Dysarthria (Nervous system disorders) | 6 | 9
Dysgeusia (Nervous system disorders) | 52 | 42
Encephalopathy (Nervous system disorders) | 3 | 1
Extrapyramidal disorder (Nervous system disorders) | 0 | 1
Facial spasm (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 24 | 26
Hyperaesthesia (Nervous system disorders) | 1 | 0
Hypersomnia (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 6 | 5
Intellectual disability (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 4 | 3
Mental impairment (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 1 | 0
Muscle contractions involuntary (Nervous system disorders) | 1 | 0
Muscle spasticity (Nervous system disorders) | 1 | 2
Myoclonus (Nervous system disorders) | 0 | 1
Nervous system disorder (Nervous system disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 1 | 2
Neuropathy peripheral (Nervous system disorders) | 105 | 80
Neurotoxicity (Nervous system disorders) | 2 | 5
Paraesthesia (Nervous system disorders) | 34 | 34
Parosmia (Nervous system disorders) | 1 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 4
Peripheral sensory neuropathy (Nervous system disorders) | 55 | 60
Peroneal nerve palsy (Nervous system disorders) | 2 | 1
Polyneuropathy (Nervous system disorders) | 5 | 3
Presyncope (Nervous system disorders) | 3 | 2
Restless legs syndrome (Nervous system disorders) | 1 | 2
Sciatica (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 0 | 1
Sensory disturbance (Nervous system disorders) | 0 | 1
Sinus headache (Nervous system disorders) | 1 | 0
Sleep paralysis (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 1 | 2
Speech disorder (Nervous system disorders) | 2 | 0
Syncope (Nervous system disorders) | 10 | 4
Thermohyperaesthesia (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 6 | 6
Visual field defect (Nervous system disorders) | 1 | 0
Vocal cord paresis (Nervous system disorders) | 1 | 0
Device dislocation (Product Issues) | 1 | 0
Device malfunction (Product Issues) | 2 | 1
Device occlusion (Product Issues) | 3 | 3
Stent malfunction (Product Issues) | 1 | 2
Adjustment disorder (Psychiatric disorders) | 1 | 0
Affective disorder (Psychiatric disorders) | 0 | 1
Agitation (Psychiatric disorders) | 2 | 0
Anxiety (Psychiatric disorders) | 26 | 12
Anxiety disorder (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 3 | 2
Delirium (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 17 | 9
Disorientation (Psychiatric disorders) | 1 | 1
Drug dependence (Psychiatric disorders) | 1 | 0
Dysphoria (Psychiatric disorders) | 1 | 1
Hallucination, visual (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 36 | 30
Irritability (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 3 | 1
Panic attack (Psychiatric disorders) | 0 | 2
Paranoia (Psychiatric disorders) | 1 | 0
Restlessness (Psychiatric disorders) | 2 | 1
Sleep disorder (Psychiatric disorders) | 1 | 4
Stress (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 4 | 7
Bladder discomfort (Renal and urinary disorders) | 1 | 0
Calculus bladder (Renal and urinary disorders) | 0 | 1
Chromaturia (Renal and urinary disorders) | 3 | 2
Chronic kidney disease (Renal and urinary disorders) | 0 | 1
Cystitis noninfective (Renal and urinary disorders) | 1 | 2
Dysuria (Renal and urinary disorders) | 6 | 3
Haematuria (Renal and urinary disorders) | 3 | 4
Haemoglobinuria (Renal and urinary disorders) | 0 | 1
Micturition urgency (Renal and urinary disorders) | 4 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Nocturia (Renal and urinary disorders) | 2 | 0
Pollakiuria (Renal and urinary disorders) | 4 | 5
Polyuria (Renal and urinary disorders) | 0 | 1
Prerenal failure (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 4 | 1
Renal failure (Renal and urinary disorders) | 3 | 0
Renal pain (Renal and urinary disorders) | 1 | 0
Ureteric obstruction (Renal and urinary disorders) | 1 | 0
Urinary hesitation (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 4 | 2
Urinary retention (Renal and urinary disorders) | 5 | 5
Urinary tract pain (Renal and urinary disorders) | 2 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 2
Breast discomfort (Reproductive system and breast disorders) | 0 | 1
Breast pain (Reproductive system and breast disorders) | 1 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 1
Ovarian vein thrombosis (Reproductive system and breast disorders) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 2 | 0
Penile pain (Reproductive system and breast disorders) | 1 | 0
Scrotal oedema (Reproductive system and breast disorders) | 1 | 0
Scrotal swelling (Reproductive system and breast disorders) | 1 | 0
Testicular pain (Reproductive system and breast disorders) | 0 | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 1
Vaginal discharge (Reproductive system and breast disorders) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 1
Vulva cyst (Reproductive system and breast disorders) | 0 | 1
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 1
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 31 | 25
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 7 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 29 | 31
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Dyspnoea paroxysmal nocturnal (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 22 | 20
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 24 | 24
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 5
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 11 | 9
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 6
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 22 | 10
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 7 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 18 | 5
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 54 | 41
Blister (Skin and subcutaneous tissue disorders) | 1 | 1
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 3 | 2
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 | 5
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 17 | 7
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 2 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 | 1
Erythema (Skin and subcutaneous tissue disorders) | 6 | 6
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2 | 0
Facial wasting (Skin and subcutaneous tissue disorders) | 1 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 10 | 8
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 1
Nail discolouration (Skin and subcutaneous tissue disorders) | 3 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 1
Nail ridging (Skin and subcutaneous tissue disorders) | 1 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 7 | 4
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 | 1
Onycholysis (Skin and subcutaneous tissue disorders) | 1 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 2
Palmar erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Palmar-plantar erythrodysaesthesia (Skin and subcutaneous tissue disorders) | 15 | 7
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 | 0
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 16 | 12
Rash (Skin and subcutaneous tissue disorders) | 20 | 8
Rash erythematous (Skin and subcutaneous tissue disorders) | 3 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 | 4
Rash papular (Skin and subcutaneous tissue disorders) | 4 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 1
Rash vesicular (Skin and subcutaneous tissue disorders) | 1 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 1 | 0
Scab (Skin and subcutaneous tissue disorders) | 2 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 3 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Skin erosion (Skin and subcutaneous tissue disorders) | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 2
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 6 | 3
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 1
Skin maceration (Skin and subcutaneous tissue disorders) | 0 | 1
Skin mass (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 2
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 2
Angiopathy (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 16 | 6
Embolism (Vascular disorders) | 12 | 1
Flushing (Vascular disorders) | 7 | 1
Haematoma (Vascular disorders) | 1 | 1
Hot flush (Vascular disorders) | 1 | 1
Hypertension (Vascular disorders) | 45 | 18
Hypertensive crisis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 24 | 25
Jugular vein thrombosis (Vascular disorders) | 1 | 1
Orthostatic hypotension (Vascular disorders) | 3 | 3
Pallor (Vascular disorders) | 2 | 0
Pelvic venous thrombosis (Vascular disorders) | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0
Peripheral vascular disorder (Vascular disorders) | 1 | 0
Phlebitis (Vascular disorders) | 1 | 0
Subclavian vein thrombosis (Vascular disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 4 | 0
Thrombophlebitis superficial (Vascular disorders) | 0 | 2
Thrombosis (Vascular disorders) | 3 | 3
Varicose vein (Vascular disorders) | 1 | 0
Vena cava thrombosis (Vascular disorders) | 1 | 0
Venous thrombosis (Vascular disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-06-10): https://cdn.clinicaltrials.gov/large-docs/23/NCT03504423/Prot_002.pdf
  • Statistical Analysis Plan (2021-07-14): https://cdn.clinicaltrials.gov/large-docs/23/NCT03504423/SAP_001.pdf